CLINICAL TRIAL: NCT05730751
Title: Could Intrathecal Fentanyl Prevent Shoulder Tip Pain (STP) During and After Caesarean Section
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Adham Haggag, Associate proffesor, Ain Shams University
Other Study IDs: FMASU R213/2022
Record Dates: First submitted 2023-02-05; First posted 2023-02-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Anesthesia, Spinal; Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group F: The patients will receive 2.5 ml of hyperbaric bupivacaine 0.5 % and 25 µg fentanyl [6].
  Interventions: Procedure: spinal anesthesia; Procedure: caesarean section
- Group C: The patients will receive 2.5 ml of hyperbaric bupivacaine 0.5 %
  Interventions: Procedure: spinal anesthesia; Procedure: caesarean section

INTERVENTIONS:
Procedure: spinal anesthesia — spinal anesthesia
Procedure: caesarean section — LSCS

SUMMARY:
Shoulder pain is a commonly observed, annoying and mostly neglected consequence of cesarean section and little is known as well as explored about intraoperative shoulder pain. This study will explore the factors precipitating shoulder pain during cesarean section, preventive analgesia and treatment modalities

DETAILED DESCRIPTION:
The most common surgery performed on women around the world is caesarean section. The majority of caesarean sections these days are carried out under regional analgesia, though some need to be carried out under general anesthesia, particularly in emergency situations or when there is a contraindication to the use of regional anesthesia. Benefits of spinal anesthesia include an awake mother at birth, minimizing or avoiding the risk of general anesthesia (aspiration, difficulty intubation, etc.) and minimal side effects to the newborn.

Shoulder tip pain (STP) is a usual complication after laparoscopy with the incidence reported varying between35% to 80%. Recent studies suggest that this type of pain is also seen after cesarean section Shoulder pain is commonly observed, but is largely ignored complication of caesarean section, and little is understood or studied regarding intraoperative shoulder pain.

Shoulder pain can be more excruciating in some patients than the pain from the surgical incision. This pain may be associated with diaphragmatic irritation/injury from local acidosis, the irritating effects of carbon dioxide during pneumoperitoneum, or stretching forces on the diaphragm. ( Although carbon dioxide is not used in cesarean compared to laparoscopic surgeries, stretching forces on the diaphragm during cesarean can be one of the causes of shoulder pain in these patients.

It is believed that seepage of blood or amniotic fluid into the abdomen accumulation during cesarean section and subdiaphragmatic may be the cause of STP. Retained blood clots in patients undergoing CS can induce diaphragmatic discomfort and stimulate the phrenic nerve. Peritoneal cleaning and visceral manipulation also may play a part.

Fentanyl is a commonly used lipophilic opioid for spinal anesthesia with relatively approved intraoperative anti-nociceptors effect.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II,
* uncomplicated, singleton pregnancies of at least 36 weeks gestation.

Exclusion Criteria:

* Cardiac, liver or renal disease
* Allergy to amide local anesthetics
* History of epilepsy or any other neurological problem
* Any contraindication of regional anesthesia, or patient refusal
* Intrauterine growth restriction or fetal compromise

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: parturients undergoing LSCS
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
incidence of occurrence intraoperative and early postoperative shoulder tip pain anesthesia as a preventive analgesia for shoulder tips pain with Cesarean section. | intraoperative till 12 hours postoperative
  comparing incidence of shoulder pain between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt